CLINICAL TRIAL: NCT06341413
Title: Sleep and Emotion Processing in Adolescent Post-Traumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1281; A539500 (Other: UW- Madison); SMPH/SLEEP CENTER/SLEEP CTR (Other: UW- Madison); Protocol Approved 8/6/2024 (Other: UW- Madison); 1R01MH132221 (NIH)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation mode first (Experimental): During one week, the SmartSleep device will be set to stimulation mode.
  Interventions: Device: SmartSleep device
- Sham mode first (Sham Comparator): During one week, the SmartSleep device will be set to sham.
  Interventions: Device: SmartSleep device

INTERVENTIONS:
Device: SmartSleep device — Device worn during sleep

SUMMARY:
The goal of this clinical trial is to characterize the role of sleep, emotion processing, and daily affect in post-traumatic stress disorder (PTSD) and whether improving sleep quality using slow wave activity enhancement will impact next-day affect in youth.

Participants will attend 4 study visits:

* A clinical and trauma assessment visit
* A testing day that may include cognitive testing, surveys, and an MRI.
* An overnight sleep study following one week of at-home sleep recordings with the device in the sham condition
* An overnight sleep study following one week of at-home sleep recordings with the device in the sleep enhancement condition

DETAILED DESCRIPTION:
In this study, researchers aim to characterize sleep and explore its relationship to emotion processing and daily affect in 165 youth spilt into 3 groups. Researchers will use advanced sleep assessment methodologies including: (1) high-density EEG (256 channels) in the laboratory to explore the regional distribution of sleep before and after an emotional learning task and; (2) a sleep-wearable EEG recording headband, SmartSleep, to record sleep longitudinally at home. Using SmartSleep's sleep enhancement algorithms, researchers will determine whether the deepest sleep, slow-wave activity (SWA) of non-rapid eye-movement (NREM) sleep, can be reliably increased in all youth.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the following criteria:

* Aged 15-18 years old, inclusive
* Must agree to inform the investigators within 48 hours of any emergent medical conditions and procedures
* Able to lie still on their back for up to 1 hour
* Must not be pregnant
* Must agree not to participate in any other interventional clinical trials during the duration of the study
* Must be willing to comply with all study procedures
* Agree to have study visits video and/or audio recorded, including consent visit, clinical assessments (for staff training) and in-laboratory sleep visits (recording deleted within one month of study visit).
* A primary parent or guardian is willing participate in the study and to provide informed consent
* Are fluent in or predominantly speaking and reading in English

In addition, PTSD and TEC youth must satisfy the following criteria:

- Must have a history of at least one traumatic event of any type, as defined by the DSM-V. This may include exposure to physical or sexual abuse, witnessing violence against loved ones or friends, traumatic accidents, natural disasters, death of a close family member etc.

Additional criteria for PTSD youth:

- At baseline, meet threshold for DSM-5 criteria for current severe PTSD, as determined by the semi-structured clinical interview (KSADS).

Exclusion Criteria:

* Caregiver or adolescent is unwilling or unable to give adequate informed consent.
* Are likely, in the investigator's opinion and via observation during the screening and clinical assessment period, to be re-exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation during study participation.
* Any finding(s), based on the screening process, that the PI feels would make the study unsuitable for the participant.
* Participation in the last 30 days in a clinical study involving an investigational drug
* MRI contraindication
* Claustrophobia or inability lie still in the scanner after practice MRI sessions.
* Any participant presenting current serious suicide risk, as determined through the KSADS, responses to C-SSRS, and/or clinical judgment of the investigator, will be excluded; however, history of suicide attempts is not an exclusion. Would present a serious risk to others as established through clinical interview and contact with treating physician.
* Neurodevelopmental disorders such as autism spectrum disorder
* Intellectual Disability (IQ less than 70, per self-report)
* Currently impaired by any medical condition that would prevent study participation
* Traumatic brain injury with ongoing symptoms, including headache, visual disturbances, and/or impairments in concentration.
* Neurological disorder(s) such as seizures, epilepsy, or brain tumors (Tourette's disorder, as diagnosed in the KSADS, is not exclusionary for TEC/PTSD youth)
* Current use of medications or other drugs (i.e., alcohol) in a manner that may interfere with sleep.
* Possible pregnancy

Exclusions for Typically developing youth:

* No history of or current psychopathology, as defined in the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS), with exception of past specific phobia.
* Current diagnosis of a sleep disorder (self-report).
* Any history of any traumatic experience as defined by the DSM-V, including IPV exposure, neglect, or emotional abuse etc.

PTSD Youth:

- Current diagnosis of or history of psychotic disorder, bipolar disorder, or autism spectrum disorder diagnosed by the KSADS interview. No other co-morbid disorders are exclusionary.

TEC Youth:

- A current diagnosis of PTSD or a current diagnosis of or history of psychotic disorder, bipolar disorder, or autism spectrum disorder diagnosed by the KSADS interview.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Regulation - arousal | First overnight session to second overnight, up to 5 weeks
  Participants will view 140 target stimuli - 70 negative and 70 neutral- in pseudorandom order. The Self-Assessment Manikin Scale for Arousal 142 (SAM) appears after the target image and participants are asked to rate degree of emotional arousal experienced while processing the picture by pressing one of nine response buttons (ranging from 1 = very low to 9 = very high).
Change in Emotional Regulation - recall | First overnight session to second overnight, up to 5 weeks
  Participants complete a recognition phase. In this phase, 200 neutral and negative images are viewed. This set includes the 140 previously viewed images intermixed with 70 novel images (50% negative and 50% neutral). Participants are asked to assess arousal using the SAM (degree of emotional arousal experienced while processing the picture by pressing one of nine response buttons (ranging from 1 = very low to 9 = very high)), and to indicate whether or not they recognize pictures from the previous encoding session (''old'') or not (''new'') by pressing one of two response buttons.
Change in Slow-wave Activity (SWA) | First overnight session to second overnight, up to 5 weeks
  Measured by overnight high-density EEG

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) | First week at-home recordings to second week, up to 6 weeks
  PANAS consists of 10 positive and 10 negative valence word items. Items are rated by the participant to indicate their assessment of how they are feeling about this item "right now" on a scale of 1(slightly) or not at all through 5 (extremely). 10 of of the items form a positive affect subscale, in which a higher score indicates increased positive affect, with a subscale range of 10 to 50. 10 of the items form a negative affect subscale, in which a higher score indicates more negative affect, with a subscale range of 10 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Jones, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No